CLINICAL TRIAL: NCT01423773
Title: Ocular Comfort and OCT Observation of Post Lens Clearance and Ocular Tissue Compression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CIBA VISION (Industry)
Collaborators: Bascom Palmer Eye Institute (Other)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: P-367-C-800
Record Dates: First submitted 2011-08-25; First posted 2011-08-26 (Estimated); Results first posted 2012-12-21 (Estimated); Last update posted 2013-06-28 (Estimated); Status verified 2012-11

CONDITIONS: Ocular Comfort

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lotrafilcon A test/lotrafilcon A control (Other): Lotrafilcon A test contact lens worn first, with lotrafilcon A control contact lens worn second. Each product worn bilaterally for two days as follows: 20 minutes on Day 1 and 10 hours on Day 2.
  Interventions: Device: Lotrafilcon A test contact lens; Device: Lotrafilcon A control contact lens; Device: Ultra-High Resolution Optical Coherence Tomographer (OCT)
- Lotrafilcon A control/lotrafilcon A test (Other): Lotrafilcon A control contact lens worn first, with lotrafilcon A test contact lens worn second. Each product worn bilaterally for two days as follows: 20 minutes on Day 1 and 10 hours on Day 2.
  Interventions: Device: Lotrafilcon A test contact lens; Device: Lotrafilcon A control contact lens; Device: Ultra-High Resolution Optical Coherence Tomographer (OCT)

INTERVENTIONS:
Device: Lotrafilcon A test contact lens — Silicone hydrogel single vision, soft contact lens with alternate parameters
Device: Lotrafilcon A control contact lens — Silicone hydrogel single vision, soft contact lens
  Other Names: Night&Day
Device: Ultra-High Resolution Optical Coherence Tomographer (OCT) — Investigational, nonsignificant risk device for measuring post lens clearance and ocular tissue compression during contact lens wear

SUMMARY:
The purpose of this study was to compare the fit and comfort of two types of contact lenses.

DETAILED DESCRIPTION:
The relationship between ocular comfort and the Optical Coherence Tomography (OCT) measurements of post lens clearance and ocular tissue compression was studied.

ELIGIBILITY:
Inclusion Criteria:

* Be of legal age of consent and sign Informed Consent document.
* Normal binocularity.
* Be able to wear soft contact lenses.
* Willing to comply with the wear and study visit schedule.
* Spherical contact lens prescription within 0.50 diopter of the available lens powers.
* Spectacle cylinder less than or equal to 1.50 diopter.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Eye injury or surgery within twelve weeks of enrollment.
* Pre-existing ocular irritation that would preclude contact lens fitting.
* Currently enrolled in any clinical trial.
* Evidence of systemic or ocular abnormality, infection, or disease likely to affect successful wear of contact lenses or use of accessory solutions as determined by the investigator.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jianhua Wang, MD, PhD, Principal Investigator — Bascom Palmer Eye Institute
Locations (1):
- McKnight Building, Bascom Palmer Eye Institute, Miami, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Partipants were recruited from one US study center.
Pre-assignment Details: This reporting group includes all enrolled participants.
Groups:
- Lotrafilcon A Test, Then Lotrafilcon A Control: Lotrafilcon A test contact lenses worn in Period One, with lotrafilcon A control contact lenses worn in Period Two. Each product was worn bilaterally for two consecutive days as follows: 20 minutes on Day 1, and 10 hours on Day 2. A wash-out of 24 hours minimum to 3 weeks maximum separated the two periods.
- Lotrafilcon A Control, Then Lotrafilcon A Test: Lotrafilcon A control contact lenses worn in Period One, with lotrafilcon A test contact lenses worn in Period Two. Each product was worn bilaterally for two consecutive days as follows: 20 minutes on Day 1, and 10 hours on Day 2. A wash-out of 24 hours minimum to 3 weeks maximum separated the two periods.
Period: Period One, 2 Days
Arm/Group | Lotrafilcon A Test, Then Lotrafilcon A Control | Lotrafilcon A Control, Then Lotrafilcon A Test
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Period 2, 2 Days
Arm/Group | Lotrafilcon A Test, Then Lotrafilcon A Control | Lotrafilcon A Control, Then Lotrafilcon A Test
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall: Each product worn bilaterally for two consecutive days in either Period One or Period Two. A wash-out of 24 hours minimum to 3 weeks maximum separated the two periods.
Arm/Group | Overall
Number analyzed (Participants) | 20
Age Continuous [Mean (Standard Deviation); unit: years] | 36.0 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Final Comfort
Description: Comfort was assessed by the participant on a Visual Analog Scale of 0 to 100, where 0=Extremely Uncomfortable ("My eyes are in pain. I cannot tolerate my lenses") and 100=Extremely Comfortable ("My eyes feel GREAT, better than normal. I cannot feel my lenses").
Time Frame: Day 2, Hour 10
Population: All enrolled participants
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Lotrafilcon A Test: Lotrafilcon A test contact lenses worn for two consecutive days as follows: 20 minutes on Day 1, and 10 hours on Day 2.
- Lotrafilcon A Control: Lotrafilcon A control contact lenses worn for two consecutive days as follows: 20 minutes on Day 1, and 10 hours on Day 2.
Arm/Group | Lotrafilcon A Test | Lotrafilcon A Control
Number analyzed (Participants) | 20 | 20
Units on a scale | 87.6 (10.5) | 87.9 (11.1)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study.
Description: This reporting group includes all enrolled participants.
Arm/Group | Lotrafilcon A Test | Lotrafilcon A Control
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

LIMITATIONS AND CAVEATS:
The sample size may be small for establishing relationship between ocular comfort and other measurable variables.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No